CLINICAL TRIAL: NCT02121015
Title: Online Collaborative Learning Intervention to Prevent Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Northwestern University (Other); University of Iowa (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Duffecy, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-1181; 1R34MH102478-01 (NIH); 7R34MH102478-02 (NIH)
Record Dates: First submitted 2014-02-17; First posted 2014-04-23 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Depression, Postpartum
Keywords: Postpartum Depression; Depression Prevention; Supportive Accountability; Individual Internet Interventions (IIIs); Internet Support Groups (ISGs)
MeSH Terms: conditions — Depression, Postpartum | interventions — Reimbursement, Disproportionate Share

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Self-Directed (Active Comparator): Access to the e-health intervention (an interactive website with didactic material and interactive tools) for participants to use at their own pace for 8 weeks (Self-Directed)
  Interventions: Behavioral: Self-Directed
- Share (Experimental): Access to the same e-health intervention + an internet social networking component consisting of up to 12 other pregnant women (Share).
  Interventions: Behavioral: Share

INTERVENTIONS:
Behavioral: Share
  Arms: Share
Behavioral: Self-Directed
  Arms: Self-Directed

SUMMARY:
The overarching aim of this project is to develop and pilot an innovative online intervention (Share) that integrates an Individual Internet Intervention (III) and an Internet Support Group (ISG) in preventing Postpartum Major Depression (PPMD). To establish that supportive accountability is a critical component of the intervention, Share will be compared to an III alone, and an ISG without the III components.

DETAILED DESCRIPTION:
Postpartum major depression (PPMD) occurs in approximately 7% of women in the first three months after childbirth and up to 22% of women over the first year postpartum. The impact of PPMD can be profound, including emotional distress, impairment in daily functioning and especially in caring for an infant for women as well as disturbances in infant development. The need for preventive interventions that are effective and widely accessible is clear and widely recognized.

While several psychological interventions to prevent PPMD have demonstrated efficacy, all of these interventions require women to be physically present at a treatment site at a particular time and day. There are numerous well established access barriers to traditional face-to-face psychological interventions, particularly for postpartum women facing the demands of childcare, including cost, transportation barriers, and time constraints, all of which make it impossible for the vast majority of women to participate in preventive care. The Internet offers great potential in extending mental health services to perinatal women because it directly circumvents these barriers.

Two broad classes of internet interventions have been evaluated within medicine generally, although to date there are no published evaluations of such interventions among perinatal women: Individual Internet Interventions (IIIs), which provide patients with access to web-based self-management programs, and Internet Support Groups (ISGs), which are usually centered around a discussion board or chat room. Meta-analyses suggest that IIIs are effective with acutely depressed patients when they include regular support by live coach (d=.61), but are much less effective when they are provided as a stand-alone treatment (d=.25). The enhanced efficacy of coach-supported IIIs appears to be due to the greater adherence to the intervention (e.g. more frequent usage) resulting from personal coach contact. The obvious drawbacks are cost and scalability: infrastructures for the training, oversight and payment of coaches must be implemented.

In contrast, ISGs provide a vehicle for peer support, and are very highly valued and commonly used by perinatal women. However, while adherence may be good, trials have found unmoderated ISGs to be ineffective at reducing distress and depression, Taken together, the efficacy of the IIIs and the adherence, flexibility, and potential for peer support in an ISG suggest that peers in a well-constructed ISG that encourages support and collaborative learning, could enhance adherence and outcomes of online self-management training programs. Learning these self-management skills have proven effective in face-to-face interventions to prevent depression among perinatal women.

This intervention, which we call "Share", is based upon a unique combination of two critical concepts:

1. the capacity of IIIs to teach self-management skills; and
2. the potential for ISGs to enhance adherence and contribute to effective learning.

ELIGIBILITY:
Inclusion Criteria:

Women who are:

1. 18 years and older
2. Pregnant and between 20 and 28 weeks gestation and for whom there is an expectation of a full 40 week gestation at the birth of their child
3. Have a Patient Health Questionnaire (PHQ-9) score score between 5-14
4. Have access to a broadband internet connection
5. Are able to read and speak English

Exclusion Criteria:

Women who:

1. Have visual, hearing, voice, or motor impairment that would prevent completion of study procedures
2. Are diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, substance use disorder or other diagnosis using the Mini International Neuropsychiatric Interview (MINI) for which participation in this trial is either inappropriate or dangerous
3. Are currently receiving treatment (medication or psychotherapy), or have an intention to resume antidepressant medication after delivery (i.e., women who discontinued their medication during pregnancy)
4. Are suicidal (i.e., have ideation, plan, and intent)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in depression symptoms over time as measured by the Inventory of Depression and Anxiety Symptoms (IDAS) | Week 20

SECONDARY OUTCOMES:
Usability and satisfaction based on the USE measure | Week 20
Diagnosis of Major Depressive Disorder based on the Mini International Neuropsychiatric Interview (MINI) | Week 20
Site usage as measured by the number of logins to the site over the course of the intervention | Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Duffecy, PhD, Principal Investigator — University of Illinois at Chicago
Locations (3):
- United States (3):
  - University of Illinois at Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa

REFERENCES:
- [Derived] Duffecy J, Grekin R, Long JD, Mills JA, O'Hara M. Randomized controlled trial of Sunnyside: Individual versus group-based online interventions to prevent postpartum depression. J Affect Disord. 2022 Aug 15;311:538-547. doi: 10.1016/j.jad.2022.05.123. Epub 2022 May 30. PMID 35654284
- [Derived] Duffecy J, Grekin R, Hinkel H, Gallivan N, Nelson G, O'Hara MW. A Group-Based Online Intervention to Prevent Postpartum Depression (Sunnyside): Feasibility Randomized Controlled Trial. JMIR Ment Health. 2019 May 28;6(5):e10778. doi: 10.2196/10778. PMID 31140443